CLINICAL TRIAL: NCT06137664
Title: A Phase 1/2, Randomized, Observer-Blind, Active-Controlled, Age De-escalation, Dose Combination Ranging Study to Assess the Safety and Immunogenicity of Co-administered Novel Live Attenuated Trivalent Oral Poliomyelitis Vaccine in Healthy Adults, Young Children, and Neonates and Co-administered Novel Live Attenuated Monovalent Oral Poliomyelitis Vaccines 1 and 2 in Neonates in Bangladesh
Brief Title: Study of Trivalent and Bivalent (Types 1 & 2) Novel Oral Poliomyelitis Vaccines
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Bio Farma, Indonesia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CVIA 095
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Poliomyelitis
Keywords: poliovirus vaccine; Trivalent oral poliovirus vaccine; Novel oral poliovirus vaccine
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- Adults: High-dose (HD) nOPV1 + HD nOPV2 + HD nOPV3 (Experimental): Adults will receive nOPV1 (10^6.5 Cell Culture Infectious Dose 50% [CCID₅₀]) plus nOPV2 (10^5.6 CCID₅₀) plus nOPV3 (10^6.5 CCID₅₀) on Day 1 and Day 29.
  Interventions: Biological: Novel oral poliomyelitis vaccine type 1 (nOPV1); Biological: Novel oral poliomyelitis vaccine type 2 (nOPV2); Biological: Novel oral poliomyelitis vaccine type 3 (nOPV3)
- Adults:bOPV (Active Comparator): Adults will receive bivalent OPV (types 1 and 3) on Day 1 and Day 29. Each dose (2 drops = 0.1 mL) contains >10^6.0 infective units of type 1 and >10^5.8 of type 3.
  Interventions: Biological: Bivalent Oral Poliomyelitis Vaccine (bOPV)
- Young Children: Middle-dose (MD) nOPV1 + Low-dose (LD) nOPV2 + MD nOPV3 (Experimental): Children aged ≥ 1 to < 5 years old will receive nOPV1 (10^6.0 CCID₅₀) plus nOPV2 (10^5.3 CCID₅₀) plus nOPV3 (10^6.0 CCID₅₀) on Day 1 and Day 29.
  Interventions: Biological: Novel oral poliomyelitis vaccine type 1 (nOPV1); Biological: Novel oral poliomyelitis vaccine type 2 (nOPV2); Biological: Novel oral poliomyelitis vaccine type 3 (nOPV3)
- Young Children: HD nOPV1 + HD nOPV2 + HD nOPV3 (Experimental): Children aged ≥ 1 to < 5 years old will receive nOPV1 (10^6.5 CCID₅₀) plus nOPV2 (10^5.6 CCID₅₀) plus nOPV3 (10^6.5 CCID₅₀) on Day 1 and Day 29.
  Interventions: Biological: Novel oral poliomyelitis vaccine type 1 (nOPV1); Biological: Novel oral poliomyelitis vaccine type 2 (nOPV2); Biological: Novel oral poliomyelitis vaccine type 3 (nOPV3)
- Young Children: Low-dose (LD) nOPV2 (Active Comparator): Children aged ≥ 1 to < 5 years old will receive nOPV2 (10^5.3 CCID₅₀) on Day 1 and Day 29.
  Interventions: Biological: Novel oral poliomyelitis vaccine type 2 (nOPV2)
- Young Children: bOPV (Active Comparator): Children aged ≥ 1 to < 5 years old will receive bivalent OPV (types 1 and 3) on Day 1 and Day 29. Each dose (2 drops = 0.1 mL) contains > 10^6.0 infective units of type 1 and > 10^5.8 of type 3.
  Interventions: Biological: Bivalent Oral Poliomyelitis Vaccine (bOPV)
- Neonates: MD nOPV1 + LD nOPV2 + MD nOPV3 (Experimental): Newborns will receive nOPV1 (10^6.0 CCID₅₀) plus nOPV2 (10^5.3 CCID₅₀) plus nOPV3 (10^6.0 CCID₅₀) at birth, week 6, week 10 and week 14 of life.
  Interventions: Biological: Novel oral poliomyelitis vaccine type 1 (nOPV1); Biological: Novel oral poliomyelitis vaccine type 2 (nOPV2); Biological: Novel oral poliomyelitis vaccine type 3 (nOPV3)
- Neonates: HD nOPV1 + LD nOPV2 + HD nOPV3 (Experimental): Newborns will receive nOPV1 (10^6.5 CCID₅₀) plus nOPV2 (10^5.3 CCID₅₀) plus nOPV3 (10^6.5 CCID₅₀) at birth, week 6, week 10 and week 14 of life.
  Interventions: Biological: Novel oral poliomyelitis vaccine type 1 (nOPV1); Biological: Novel oral poliomyelitis vaccine type 2 (nOPV2); Biological: Novel oral poliomyelitis vaccine type 3 (nOPV3)
- Neonates: MD nOPV1 + LD nOPV2 + HD nOPV3 (Experimental): Newborns will receive nOPV1 (10^6.0 CCID₅₀) plus nOPV2 (10^5.3 CCID₅₀) plus nOPV3 (10^6.5 CCID₅₀) at birth, week 6, week 10 and week 14 of life.
  Interventions: Biological: Novel oral poliomyelitis vaccine type 1 (nOPV1); Biological: Novel oral poliomyelitis vaccine type 2 (nOPV2); Biological: Novel oral poliomyelitis vaccine type 3 (nOPV3)
- Neonates: HD nOPV1+ LD nOPV2+ MD nOPV3 (Experimental): Newborns will receive nOPV1 (10^6.5 CCID₅₀) plus nOPV2 (10^5.3 CCID₅₀) plus nOPV3 (10^6.0 CCID₅₀) at birth, week 6, week 10 and week 14 of life.
  Interventions: Biological: Novel oral poliomyelitis vaccine type 1 (nOPV1); Biological: Novel oral poliomyelitis vaccine type 2 (nOPV2); Biological: Novel oral poliomyelitis vaccine type 3 (nOPV3)
- Neonates: HD nOPV1 + HD nOPV2 + HD nOPV3 (Experimental): Newborns will receive nOPV1 (10^6.5 CCID₅₀) plus nOPV2 (10^5.6 CCID₅₀) plus nOPV3 (10^6.5 CCID₅₀) at birth, week 6, week 10 and week 14 of life.
  Interventions: Biological: Novel oral poliomyelitis vaccine type 1 (nOPV1); Biological: Novel oral poliomyelitis vaccine type 2 (nOPV2); Biological: Novel oral poliomyelitis vaccine type 3 (nOPV3)
- Neonates: bOPV (Active Comparator): Newborns will receive bivalent OPV (types 1 and 3) at birth, week 6, week 10 and week 14 of life. Each dose (2 drops = 0.1 mL) contains >10^6.0 infective units of type 1 and >10^5.8 of type 3.
  Interventions: Biological: Bivalent Oral Poliomyelitis Vaccine (bOPV)
- Neonates: MD nOPV1 + LD nOPV2 (Experimental): Newborns will receive nOPV1 (10^6.0 CCID₅₀) plus nOPV2 (10^5.3 CCID₅₀) at birth, week 6, week 10 and week 14 of life.
  Interventions: Biological: Novel oral poliomyelitis vaccine type 1 (nOPV1); Biological: Novel oral poliomyelitis vaccine type 2 (nOPV2)
- Neonates: LD nOPV2 (Active Comparator): Newborns will receive nOPV2 (10^5.3 CCID₅₀) at birth, week 6, week 10 and week 14 of life.
  Interventions: Biological: Novel oral poliomyelitis vaccine type 2 (nOPV2)

INTERVENTIONS:
Biological: Novel oral poliomyelitis vaccine type 1 (nOPV1) — Live attenuated novel poliomyelitis virus type 1 at two different dosages, containing middle-dose (MD) 10^6.0, or high-dose (HD) 10^6.5 CCID₅₀/dose
  Arms: Adults: High-dose (HD) nOPV1 + HD nOPV2 + HD nOPV3; Neonates: HD nOPV1 + HD nOPV2 + HD nOPV3; Neonates: HD nOPV1 + LD nOPV2 + HD nOPV3; Neonates: HD nOPV1+ LD nOPV2+ MD nOPV3; Neonates: MD nOPV1 + LD nOPV2; Neonates: MD nOPV1 + LD nOPV2 + HD nOPV3; Neonates: MD nOPV1 + LD nOPV2 + MD nOPV3; Young Children: HD nOPV1 + HD nOPV2 + HD nOPV3; Young Children: Middle-dose (MD) nOPV1 + Low-dose (LD) nOPV2 + MD nOPV3
Biological: Novel oral poliomyelitis vaccine type 2 (nOPV2) — Live attenuated novel poliomyelitis virus type 2 administered at low-dose (LD) 10^5.3 and HD 10^5.6 CCID₅₀/dose.
  Arms: Adults: High-dose (HD) nOPV1 + HD nOPV2 + HD nOPV3; Neonates: HD nOPV1 + HD nOPV2 + HD nOPV3; Neonates: HD nOPV1 + LD nOPV2 + HD nOPV3; Neonates: HD nOPV1+ LD nOPV2+ MD nOPV3; Neonates: LD nOPV2; Neonates: MD nOPV1 + LD nOPV2; Neonates: MD nOPV1 + LD nOPV2 + HD nOPV3; Neonates: MD nOPV1 + LD nOPV2 + MD nOPV3; Young Children: HD nOPV1 + HD nOPV2 + HD nOPV3; Young Children: Low-dose (LD) nOPV2; Young Children: Middle-dose (MD) nOPV1 + Low-dose (LD) nOPV2 + MD nOPV3
Biological: Novel oral poliomyelitis vaccine type 3 (nOPV3) — Live attenuated novel poliomyelitis virus type 3 at two different dosages, containing MD 10^6.0, or HD 10^6.5 CCID₅₀/dose.
  Arms: Adults: High-dose (HD) nOPV1 + HD nOPV2 + HD nOPV3; Neonates: HD nOPV1 + HD nOPV2 + HD nOPV3; Neonates: HD nOPV1 + LD nOPV2 + HD nOPV3; Neonates: HD nOPV1+ LD nOPV2+ MD nOPV3; Neonates: MD nOPV1 + LD nOPV2 + HD nOPV3; Neonates: MD nOPV1 + LD nOPV2 + MD nOPV3; Young Children: HD nOPV1 + HD nOPV2 + HD nOPV3; Young Children: Middle-dose (MD) nOPV1 + Low-dose (LD) nOPV2 + MD nOPV3
Biological: Bivalent Oral Poliomyelitis Vaccine (bOPV) — Live attenuated poliomyelitis viruses types 1 and 3 (Sabin strains). Each dose (2 drops = 0.1 mL) contains not less than 10^6.0 infective units of type 1 and 10^5.8 of type 3.
  Arms: Adults:bOPV; Neonates: bOPV; Young Children: bOPV

SUMMARY:
The main objectives of this study are to :

* evaluate the safety and tolerability of trivalent novel oral poliovirus vaccines (tnOPV) in healthy adults, young children, and neonates, relative to those receiving control vaccines;
* evaluate the safety and tolerability of combined novel oral poliovirus vaccine type 1 (nOPV1) + novel oral poliovirus vaccine type 2 (nOPV2) in neonates, relative to those receiving the bivalent (types 1 and 3) oral poliovirus vaccine (bOPV) control.
* compare type-specific cumulative seroconversion rates of poliovirus neutralizing antibody (NAb) titers, among all tnOPV dose combinations, following 4 vaccinations in healthy neonates;
* evaluate the type-specific cumulative seroconversion rate of poliovirus NAb titers among healthy neonates following 4 doses of combined nOPV1+nOPV2.

DETAILED DESCRIPTION:
This trial will use co-administered novel monovalent types 1, 2, and 3 vaccines to simulate administration of a potential trivalent vaccine and compare to the active control bOPV (bivalent Sabin types 1 and 3) and will be conducted at a single clinical center.

The study population will include healthy adults (≥18 to ≤45 years old) who have previously completed their full routine polio immunization series, healthy young children (≥1 to <5 years old) who have completed their full routine polio immunization series and healthy neonates (day of birth+3 days), who have not received any polio vaccination.

Enrollment in this study will be staggered into two stages and three age-descending cohorts.

Stage 1 will consist of an age-descension/dose escalation approach from adults to young children (Cohorts 1 and 2). Enrollment will begin with Cohort 1, in which 100 adults will be randomly allocated in a 1:1 ratio to Groups 1 and 2. Following a Protocol Safety Review Team (PSRT) review of the study Day 8 safety data (i.e. safety data reported up to 7 days post-vaccination #1, collected at Visit 2) of the adults in Cohort 1, and the absence of any safety concerns, 200 young children in Cohort 2 will be randomly allocated in a 1:1:1:1 ratio to Groups 3, 4, 5, and 6, respectively.

After the completion of enrollment of Cohort 2, the study will move into Stage 2. In addition to a PSRT review of Day 8 safety data of the young children in Cohort 2, there are two triggers of data from other studies to initiate the enrollment into Cohort 3:

* Absence of safety concerns upon the safety data reviews occurring at least 8 days after receipt of the first dose of 107.5 CCID50 nOPV1 or 107.5 CCID50 nOPV3 by the first 60 IPV-vaccinated infants enrolled in each of the Phase 2 monovalent trials CVIA 093 and CVIA 101, respectively (the first 45 nOPV:15 mOPV participants randomized per dose pair).
* Favorable immunogenicity data (homotypic anti-polio serum neutralizing antibody titers) from the Phase 2 monovalent nOPV1 study (CVIA 093) in IPV-vaccinated infants, and the Phase 2 monovalent nOPV3 study (CVIA 101) in young children.

Stage 2 will consist of dose exploration in neonates (Cohort 3). In Cohort 3, Groups 7-14, 2100 neonates will be randomly allocated in a 3:3:3:3:3:3:2:1 ratio, respectively.

ELIGIBILITY:
Inclusion Criteria

Inclusion Criteria for all participants:

1. Healthy, as defined by the absence of any clinically significant medical condition or congenital anomaly as determined by medical history, physical examination, and clinical assessment of the investigator.
2. Participant or parent of the participant is willing and able to provide written informed consent prior to performance of any study-specific procedure.
3. Resides and plans to remain in study area and participants and parent, when applicable, understands and is able and willing to adhere to all study visits and procedures (as evidenced by a signed informed consent form [ICF] and assessment by the investigator).

   Inclusion Criteria for Cohort 1 participants only:
4. Males or females, from 18 to 45 years of age (inclusive) at the time of enrollment.
5. If female and of childbearing potential*, not breastfeeding and not pregnant (based on a negative urine pregnancy test at screening and a negative urine pregnancy test during the 24 hours prior to any study vaccination [if screening occurs within 24 hours prior to vaccination, a single negative pregnancy test is acceptable]), agreeing to not become pregnant through other means (e.g., artificial insemination and IVF) and have repeated pregnancy tests prior to any study vaccination, and having practiced adequate contraception** for 30 days prior to first study vaccination and willing to continue using adequate contraception consistently for at least 90 days after the last study vaccination.
6. Born and raised in Bangladesh in 1990 or later; if born before 1990 or not born and raised in Bangladesh, has documentation of a complete poliomyelitis immunization series containing OPV or IPV.

   Inclusion Criteria for Cohort 2 participants only:
7. Male or female child from 1 to less than 5 years of age at the time of enrollment (from the first birthday up to the day prior to the fifth birthday).
8. Based on documentation, previously received a 3 or 4 dose primary poliomyelitis immunization series containing bOPV ± IPV, with last dose received more than 3 months prior to initial study vaccination.

   Inclusion Criteria for Cohort 3 participants only:
9. Male or female newborn neonate (day of birth+ 3-day window), at the time of initial study vaccination.
10. Prior to study vaccination has received no doses of IPV or OPV or rotavirus vaccine, based upon documentation or parental history.
11. Agreement to receive polio EPI vaccines under a modified schedule.

Exclusion Criteria

Exclusion Criteria for all participants (unless otherwise specified):

1. Presence of anyone under 10 years of age in the participant's household (living in the same house or apartment unit) who does not have complete "age appropriate" vaccination status with respect to poliovirus vaccines based on the vaccination records at the time of study vaccine administration. For household members younger than 10 years of age-appropriate vaccination is a complete series of at least three doses of OPV.
2. A known allergy, hypersensitivity, or intolerance to any components of the study vaccines, including all macrolide and aminoglycoside antibiotics (e.g., erythromycin and kanamycin).
3. Any self-reported known or suspected immunosuppressive or immunodeficiency condition (including HIV infection) in the participant or household member (living under the same roof/in the same building rather than in the same compound).
4. Receipt of any immune-modifying or immunosuppressant drugs within 6 months prior to the first study vaccine dose or planned use during the study.
5. Any known or suspected bleeding disorder in the participant that would pose a risk to venipuncture or intramuscular injection.
6. Moderate or severe (grade ≥ 2) acute illness including vomiting, diarrhea at the time of enrollment/first study vaccination - temporary exclusion.
7. Presence of fever within the 72 hours of the day of enrollment/first study vaccination (oral temperature ≥38.0˚C for Cohort 1; axillary temperature ≥37.5˚C for Cohorts 2 and 3) or any antipyretic use within past 24 hours - temporary exclusion for Cohorts 1 and 2.
8. Evidence of a clinically significant major congenital or genetic defect as judged by the investigator.
9. History of chronic administration (defined as more than 14 days) of immunosuppressant medications, including corticosteroids (> 0.5mg/kg/day or 20 mg/day of prednisolone (or equivalent) within 6 months prior to first study vaccine dose. Topical and inhaler steroids are permitted (unless indicative of a significant chronic illness otherwise excluding the young child).
10. Participation in another investigational product (drug or vaccine, including prior polio vaccine trials) clinical trial within 30 days prior to entry in this study or receipt of any such investigational product other than the study vaccine within 30 days prior to the first administration of study vaccine, or planned participation in another investigational product clinical trial during the study period.
11. Receipt of transfusion of any blood product or immunoglobulins within 12 months prior to the first administration of study vaccine or planned during the study period.
12. Participant or parent, when applicable, has any condition that in the opinion of the investigator would increase the participant's health risks in study participation or would increase the risk of not achieving the study's objectives (e.g., would compromise adherence to protocol requirements or interfere with planned safety and immunogenicity assessments).

    Exclusion Criteria for Cohort 1 participants:
13. Receipt of polio vaccine within 12 months before the start of the study.
14. Having Crohn's disease or ulcerative colitis or having had major surgery of the gastrointestinal tract involving significant loss or resection of the bowel.
15. Will have household direct or close professional contact during the study with pregnant women.
16. Will have household direct or close professional (e.g., neonatal nurses) contact during the study with children less than 2 years of age or with individuals who are encopretic (i.e., soiling of underwear with stool by children who are past the age of toilet training or other individuals, including adults, with fecal incontinence).
17. Will have professional handling of food, catering, or food production activities during the study.

    Exclusion Criteria for Cohort 2 participants:
18. Any participating children attending day care or pre-school during their participation in the study until one month after their last study vaccine administration.
19. Presence of severe malnutrition [weight-for-length/height z-score <-3SD median (per WHO published child growth standards)]-temporary exclusion if marginal and subsequently gains weight.

    Exclusion Criteria for Cohort 3 participants:
20. Low birth weight (LBW) in newborn participants which is defined as a birth weight of less than 2500 g (up to and including 2499 g) at the time of birth or by the time of enrollment
21. Premature birth (less than 37 weeks gestation).
22. From multiple birth (due to increased risk of OPV transmissions between siblings).

Ages: 0 Days to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2400 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Serious Adverse Events (SAEs) | From the time of first study vaccination through the end of the study (197 days)
  A serious adverse event is any adverse event that results in any of the following outcomes:
  1. Death.
  2. Is life-threatening.
  3. Requires inpatient hospitalization or prolongation of existing hospitalization.
  4. Results in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions.
  5. Congenital abnormality or birth defect.
  6. Important medical event that may not result in one of the above outcomes but may jeopardize the health of the study participant and require medical or surgical intervention to prevent one of the outcomes listed in the above definition of serious adverse event.
Number of Participants with Solicited Adverse Events (AEs) for 7 Days After Each Vaccination | 7 days (day of vaccination and 6 following days) after each vaccination
  Solicited AEs are pre-specified AEs that are common or known to be associated with vaccination that are actively monitored as potential indicators of vaccine reactogenicity.
Number of Participants with Unsolicited AEs for 28 Days After Each Vaccination. | 28 days (day of vaccination and 27 following days) after each vaccination
  Unsolicited AEs are any AEs reported spontaneously by the participant or parent, observed by the study personnel during study visits or identified during review of medical records or source documents.
Neonates: Seroconversion Rate of Types 1, 2, and 3 Anti-polio Serum Neutralizing Antibodies 28 Days After Last Vaccination | Baseline and 28 days following the last vaccination (week 18)
  For vaccine-naive neonates, seroconversion is defined as seropositive (titer ≥1:8) in those initially seronegative, or among those initially seropositive, as a minimum 4-fold higher (and seropositivity) than that which is expected due to maternal antibodies. This endpoint will be analyzed in neonates who receive nOPV types 1, 2, and 3.
Neonates: Seroconversion Rate of Types 1, 2, and 1 & 2 Combined Anti-polio Serum Neutralizing Antibodies 28 Days After Last Vaccination | Baseline and 28 days following the last vaccination (week 18)
  For vaccine-naive neonates, seroconversion is defined as seropositive (titer ≥1:8) in those initially seronegative, or among those initially seropositive, as a minimum 4-fold higher (and seropositivity) than that which is expected due to maternal antibodies. This endpoint will be analyzed in neonates who receive nOPV types 1 and 2 only.

SECONDARY OUTCOMES:
Neonates: Type-specific and Multitypic Seroconversion Rate of Anti-polio Serum Neutralizing Antibodies | Baseline and weeks 6, 10, 14, and 18
  For vaccine-naive neonates, seroconversion is defined as seropositive (titer ≥1:8) in those initially seronegative, or among those initially seropositive, as a minimum 4-fold higher (and seropositivity) than that which is expected due to maternal antibodies.
  Multitypic seroconversion refers to seroconversion to multiple types simultaneously, including types 1 & 2, types 1 & 3, types 2 & 3, and types 1 & 2 & 3.
Adults and Young Children: Type-specific and Multitypic Seroconversion Rate of Anti-polio Serum Neutralizing Antibodies 4 Weeks After Each Vaccination | Baseline and Weeks 4 and 8
  For previously vaccinated cohorts, seroconversion will be defined as either a minimum 4-fold rise in titer relative to the baseline value among those initially seropositive, or post-vaccination seropositivity among those seronegative at baseline.
  This endpoint will be analyzed in groups who receive nOPV types 1, 2, and 3.
All Cohorts: Types 1, 2 and 3 Anti-polio Serum Neutralizing Antibody Titers Following Last Dose | Baseline and 4 weeks following the last vaccination (week 8 in adults and young children and week 18 in neonates)
  This endpoint will be analyzed in groups who receive nOPV types 1, 2, and 3.
Adults and Young Children: Types 1, 2 and 3 Anti-polio Serum Neutralizing Antibody Titers Following First Dose | Baseline and week 4
  This endpoint will be analyzed in groups who receive nOPV types 1, 2, and 3.
All Cohorts: Geometric Mean Titer (GMT) of Types 1, 2 and 3 Anti-polio Serum Neutralizing Antibodies Following Last Dose | Baseline and 4 weeks following the last vaccination (week 8 in adults and young children and week 18 in neonates)
  This endpoint will be analyzed in groups who receive nOPV types 1, 2, and 3.
Adults and Young Children: Geometric Mean Titer (GMT) of Types 1, 2 and 3 Anti-polio Serum Neutralizing Antibodies Following First Dose | Baseline and Week 4
  This endpoint will be analyzed in groups who receive nOPV types 1, 2, and 3.
All Cohorts: Type-specific and Multitypic Seroprotection Rate Following Last Dose | Baseline and 4 weeks following the last vaccination (week 8 in adults and young children and week 18 in neonates)
  Seroprotection is defined as types 1, 2 and 3 anti-polio serum neutralizing antibody reciprocal titer ≥ 8.
  This endpoint will be analyzed in groups who receive nOPV types 1, 2, and 3.
Adults and Young Children: Type-specific and Multitypic Seroprotection Rate Following First Dose | Baseline and week 4
  Seroprotection is defined as types 1, 2 and 3 anti-polio serum neutralizing antibody reciprocal titer ≥ 8.
  This endpoint will be analyzed in groups who receive nOPV types 1, 2, and 3.
Adults and Young Children: Geometric Mean Fold Rise (GMFR) in Neutralizing Antibody Titer Relative to Previous Dose | Baseline and weeks 4 and 8
  This endpoint will be analyzed in groups who receive nOPV types 1, 2, and 3.
Neonates: Geometric Mean Fold Rise (GMFR) in Neutralizing Antibody Titer Relative to the Expected Level of Maternal Antibody and Each Pre-dose Value | Baseline and weeks 6, 10, 14, and 18
  This endpoint will be analyzed in groups who receive nOPV types 1, 2, and 3.
Neonates: Percentage of Participants Shedding Types 1, 2 and/or 3 Poliovirus Post-vaccination | From birth through 18 weeks
  Stool samples will be analyzed using polymerase chain reaction (PCR) to detect poliovirus types 1, 2, and 3.

CONTACTS AND LOCATIONS:
Locations (1):
- International Centre for Diarrhoeal Disease Research, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No